CLINICAL TRIAL: NCT02644915
Title: Effect of Edaravone on the Ischemia-Reperfusion(I/R) Injury in Kidney Transplantation Patients: A Single-Center, Double-Blinded, Randomised Controlled Trial
Brief Title: Edaravone on the Ischemia-Reperfusion(I/R) Injury in Kidney Transplantation Patients
Acronym: I/R
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xijing Hospital (Other)
Collaborators: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Principal Investigator, wangqiang, professor, Xijing Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: zxy
Record Dates: First submitted 2015-12-10; First posted 2016-01-01 (Estimated); Last update posted 2016-01-01 (Estimated); Status verified 2015-12

CONDITIONS: Kidney Transplantation
Keywords: ischemia-reperfusion(I/R) injury; Edaravone
MeSH Terms: conditions — Wounds and Injuries | interventions — Edaravone; Saline Solution

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- study group (Experimental): Edaravone 30mg dissolved in 0.9%NaCl 100ml will be treated at 10 minutes before kidney reperfusion, ending in 30 minutes.
  Standard anaesthesia and standard cure are given for all patients. During the operation we maintain the target blood pressure by keeping Central Venous Pressure(CVP)> 6 mmHg.
  Interventions: Drug: Edaravone
- control group (Placebo Comparator): 100ml 0.9%%NaCl solution,but without edaravone, will be treated at 10 minutes before kidney reperfusion, ending in 30 minutes.
  Standard anaesthesia and standard cure are given for all patients. During the operation we maintain the target blood pressure by keeping Central Venous Pressure(CVP)> 6 mmHg.
  Interventions: Drug: 0.9%%NaCl solution

INTERVENTIONS:
Drug: Edaravone — Edaravone 30mg dissolved in 0.9%NaCl 100ml will be treated at 10 minutes before kidney reperfusion , ending in 30 minutes.The number of dialysis and the serum creatinine level within the first week after the transplantation will be recorded.The participation of each patient is scheduled for 1 month.
  Other Names: Edaravone Injection
  Arms: study group
Drug: 0.9%%NaCl solution — 100ml 0.9%%NaCl solution,but without edaravone ,will be treated at 10 minutes before kidney reperfusion , ending in 30 minutes.
  Standard anaesthesia and standard cure are given for all patients. During the operation we maintain the target blood pressure by keeping Central Venous Pressure(CVP)> 6 mmHg
  Other Names: normal saline
  Arms: control group

SUMMARY:
Ischemia-reperfusion (I/R) injury is a prominent cause of delayed graft function(DGF) after kidney transplantation. Reactive oxygen species play a crucial role in I/R injury. Edaravone is a synthetic radical scavenger that has been used in acute stroke. Some animal experiments have revealed its beneficial effects against I/R injury, our goal is therefore to investigate the effectiveness of a recipient pretreatment with Edaravone at reducing the occurrence of DGF after kidney transplantation.

DETAILED DESCRIPTION:
Participants will be randomly assigned, in a 1:1 ratio, to receive Edaravone or control (0.9 %Sodium Chloride Solution,0.9%NaCl). The randomization sequence will be computer-generated, and randomization will be performed in blocks and will be stratified according to participating center.Edaravone and 0.9 %NaCl solution will be treated at 10 minutes before kidney reperfusion, ending in 30 minutes. The number of dialysis and the serum creatinine level within the first week after the transplantation will be recorded. The participation of each patient is scheduled for 1 month.

ELIGIBILITY:
Inclusion Criteria:

1. ASAⅡ-Ⅲ,elective operation patients with end-stage renal disease
2. Age 18yrs-55yrs for donors and the recipients
3. patients under hemodialysis
4. no other severe complications history for the donors and recipients
5. the first kidney transplant recipients
6. patients with written informed consent

Exclusion Criteria:

1. ASA Ⅳ
2. a second renal transplant,a multiorgan transplant or a dual kidney transplant
3. having severe comorbidity history,for example,severe cardiac dysfunction
4. cold ischemia time>24h or warm ischemia time>45min
5. variation of blood vessel ，operation time more than 2 hours
6. bleeding volume in operation>500ml and need for blood transfusion
7. participate in the other clinical trial 3 months before the enrollment
8. no suitable to participate in this experiment

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2016-03; Primary Completion 2016-09 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of DGF(postoperative complication after kidney transplantation)（%） | in the first week after the kidney transplantation
serum creatinine value (umoI/L) | within the first week

SECONDARY OUTCOMES:
average daily urinary volume（ml） | within the first week
Hospital stays after operation(d) | Participants will be followed for the duration of hospital stay, an expected average of 2 weeks
graft survival | within 30 days after surgery
other postoperative complication:acute rejection episodes、thrombosis、infections | within 30 days after surgery
Content of Malondialdehyde（mol/m l）in the blood | before transplantation and 1, 2, 3 days after transplantation
Content of Superoxide dismutase（U /m l) in the blood | before transplantation and 1, 2, 3 days after transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Qiang Wang, Study Chair — Xijing Hospital

REFERENCES:
- [Background] Zhang L, Wang F, Wang L, Wang W, Liu B, Liu J, Chen M, He Q, Liao Y, Yu X, Chen N, Zhang JE, Hu Z, Liu F, Hong D, Ma L, Liu H, Zhou X, Chen J, Pan L, Chen W, Wang W, Li X, Wang H. Prevalence of chronic kidney disease in China: a cross-sectional survey. Lancet. 2012 Mar 3;379(9818):815-22. doi: 10.1016/S0140-6736(12)60033-6. PMID 22386035
- [Background] Shah VR, Butala BP, Parikh GP, Vora KS, Parikh BK, Modi MP, Bhosale GP, Mehta T. Combined epidural and general anesthesia for paediatric renal transplantation-a single center experience. Transplant Proc. 2008 Dec;40(10):3451-4. doi: 10.1016/j.transproceed.2008.06.065. PMID 19100411
- [Background] Kontodimopoulos N, Niakas D. Overcoming inherent problems of preference-based techniques for measuring health benefits: an empirical study in the context of kidney transplantation. BMC Health Serv Res. 2006 Jan 14;6:3. doi: 10.1186/1472-6963-6-3. PMID 16412242
- [Background] Ibrahim S, Jacobs F, Zukin Y, Enriquez D, Holt D, Baldwin W 3rd, Sanfilippo F, Ratner LE. Immunohistochemical manifestations of unilateral kidney ischemia. Clin Transplant. 1996 Dec;10(6 Pt 2):646-52. PMID 8996759
- [Background] Ojo AO, Wolfe RA, Held PJ, Port FK, Schmouder RL. Delayed graft function: risk factors and implications for renal allograft survival. Transplantation. 1997 Apr 15;63(7):968-74. doi: 10.1097/00007890-199704150-00011. PMID 9112349
- [Background] Perico N, Cattaneo D, Sayegh MH, Remuzzi G. Delayed graft function in kidney transplantation. Lancet. 2004 Nov 13-19;364(9447):1814-27. doi: 10.1016/S0140-6736(04)17406-0. PMID 15541456